CLINICAL TRIAL: NCT03204708
Title: Evaluation of the Postoperative Analgesic Efficacy of Catheter Placed Interpectoral Region Via Open Technique in Patients Undergoing Modified Radical Mastectomy
Brief Title: Open Technique Interpectoral Catheter for Postoperative Analgesia in Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Guniz M.Koksal, professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 88931902-604.01.01
Record Dates: First submitted 2017-05-22; First posted 2017-07-02 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Mammary Cancer
Keywords: postoperative analgsia; peripheral block catheter; modified radical mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Catheters; Analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iv analgesia (Active Comparator): patients were given intravenously 100 mg of tramadol (contramal) 30 minutes before extubation after modified radical mastectomy.
  Interventions: Device: catheter; Drug: iv analgesia
- catheter group (Active Comparator): patients were placed a catheter under clavipectoral fascia and 30 ml of local anesthetic solution were given via catheter for postoperative analgesia
  Interventions: Device: catheter; Drug: iv analgesia

INTERVENTIONS:
Device: catheter — catheter was placed under clavipectoral fascia by open technique by surgeon at the 1/3 lateral part of clavicula neighbourhood of nervus thoracicus longus, nervus thoracodorsalis, nervus pectoralis lateralis, nervus pectoralis medialis
Drug: iv analgesia — patients were given 100 ml of tramadol 30 minutes before extubation

SUMMARY:
patients undergoing modified radical mastectomy were divided into two groups. patients in catheter group were placed a catheter with open technique by the surgeon in the pectoral area. thirty minutes before extubation %1 lidocain 10 ml, %0.5 bupivacain 10 ml and 10 ml %0.9 sodium chloride were given through the catheter for postoperative analgesia. patients in iv analgesia group were given 100 mg tramadol iv 30 minutes before extubation. visual analog pain scale (VAS) scores, rescue analgesic requirement, complications were recorded and compared between two groups 1, 6, 12, 24 hours and 90 days after surgery.

DETAILED DESCRIPTION:
patients undergoing modified radical mastectomy were divided into two groups by computer. patients in catheter group were placed a catheter under clavipectoral fascia in the neighbourhood of nervus thoracicus longus, nervus thoracodorsalis, nervus pectoralis lateralis, nervus pectoralis medialis at the 1/3 lateral part of clavicula. solution included 10 ml of %0.5 bupivacain, %1 lidocain, 10 ml %0.9 sodium chloride totally 30 ml were given via the catheter for postoperative analgesia at the end of surgery. patients in iv analgesia group were given 100 mg tramadol iv 30 minutes before extubation. Patients in both groups were given dexketoprofen 50 mg iv if the VAS score was over 4. VAS scores, rescue analgesic requirement and timing, complications were recorded and compared between groups 1, 6, 12, 24 hours and 90 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Americans Class I-II

Exclusion Criteria:

* male
* allergy to local anesthetics or
* anticoagulant drug use
* central or peripheric nerve disease
* pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — breast cancer
Enrollment: 86 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
VAS scores | 1 hour after operation
  patients were asked to give a point between 0 to 10 for their pain level. 0 is no pain, 10 is the strongest pain.
VAS scores | 6 hours after operation
  patients were asked to give a point between 0 to 10 for their pain level. 0 is no pain, 10 is the strongest pain.
VAS scores | 12 hours after operation
  patients were asked to give a point between 0 to 10 for their pain level. 0 is no pain, 10 is the strongest pain.
VAS scores | 24 hours after operation
  patients were asked to give a point between 0 to 10 for their pain level. 0 is no pain, 10 is the strongest pain.

SECONDARY OUTCOMES:
VAS scores | 3 months after operation
  patients were asked to give a point between 0 to 10 for their pain level. 0 is no pain, 10 is the strongest pain.

OTHER OUTCOMES:
rescue analgesic requirement | 1, 6, 12 and 24 hours after operation
  patients whose VAS scores were over 4 were given 50 mg of dexketoprofen in Group I, 10 ml %0.25 bupivacain in Group II

CONTACTS AND LOCATIONS:
Overall Officials: cigdem akyol beyoglu, MD, Study Director — Istanbul University

IPD SHARING:
Plan to Share IPD: No